CLINICAL TRIAL: NCT05919888
Title: SURGX Antimicrobial Gel Versus Povidone-iodine Skin Incision Prep for the Prevention of Bacterial Seeding in Total Shoulder Arthroplasty
Brief Title: SURGX Antimicrobial Gel Versus Povidone-iodine Skin Incision Prep in Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Next Science LLC (Unknown)
Responsible Party: Principal Investigator, Randall J. Otto, MD, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 32325
Record Dates: First submitted 2023-06-01; First posted 2023-06-26 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Surgery; Surgical Site Infection; Cutibacterium Acnes; Prosthetic-joint Infection
Keywords: Antimicrobial wound gel; SURGX; Betadine; Dermal layer; Skin preparation
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical trial in which patients will be assigned a study arm in sequential fashion.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- No skin incision preparation (No Intervention): All patients will receive standard pre-operative prophylactic antibiotics. Participants will all receive the same preoperative external skin preparation with Hibiclens (chlorhexidine) and ChloraPrep (2% chlorhexidine gluconate / 70% isopropyl alcohol solution) prior to draping. Intra-operative irrigation will be standardized with Irrisept (chlorhexidine gluconate 0.05% in sterile water).
  The control group will receive no dermal layer skin preparation. At the time of the surgery, after the skin incision has been made with a skin knife, the dermal layer will not be prepped with an agent.
- Povidone-iodine (Active Comparator): At the time of the surgery, after the skin incision has been made, the dermal layer be prepped with povidone-iodine.
  Drug: povidone-iodine Dose: swabstick Administration: swab the incision Frequency: once
  Interventions: Drug: Povidone-Iodine
- SURGX Wound Gel (Experimental): At the time of the surgery, after the skin incision has been made, the dermal layer be prepped with SURGX Wound Gel. SURGX wound gel is a topical antiseptic gel agent to be used on surgical incisions to prevent bacterial infection.
  Interventions: Device: SURGX Wound Gel

INTERVENTIONS:
Drug: Povidone-Iodine — Applied to skin incision.
  Other Names: Betadine
  Arms: Povidone-iodine
Device: SURGX Wound Gel — Applied to skin incision.
  Arms: SURGX Wound Gel

SUMMARY:
Comparing the growth of intra-operative tissue cultures of Cutibacterium Acnes after primary shoulder replacement when using a no-prep control group versus antimicrobial wound gel versus betadine applied to the skin layer after the skin incision has been made. Reducing the bacteria present in the deep tissues at the end of the surgery may prevent infections from developing in the future.

DETAILED DESCRIPTION:
Cutibacterium acnes (C. acnes) prosthetic joint infection is a devastating and somewhat unique complication to shoulder arthroplasty. It is a very slow-growing, aerotolerant anaerobic, non-spore forming, gram-positive rod-shaped bacteria that takes up to 2-3 weeks to grow in a lab setting. There have been several studies assessing various agents in the fight to prevent C. acnes prosthetic joint infection. These agents include standard peri-operative measures typically taken when performing shoulder replacement surgery - pre-operative prophylactic antibiotics, pre-operative skin cleanse/wash, topical adjuvants (povidone-iodine, chlorhexidine, etc.), and intra-operative antibiotic powders. The overall infection rate of shoulder arthroplasty has been cited to be between 0.9-2.9%, with C. acnes being the most common bacterium in shoulder arthroplasty periprosthetic infections. Morbidity and cost associated with shoulder prosthetic joint infection is extremely high, requiring multiple surgeries and months of treatment to overcome the infection.

One of the main issues with C. acnes is its preferred location within the body, residing within the sebaceous glands of the hair follicles, deep to the epidermis where many preoperative topical preparations to cleanse the skin prior to surgery have little affect. These glands are commonly found around the shoulder and upper back, and lead to acne. C. acnes, along with other common prosthetic joint infection bacteria, quickly create a biofilm which is impenetrable to most antibiotic agents, further stressing the importance of prevention. Recently there have been studies analyzing the effects of Benzoyl Peroxide (BPO) on C. acnes as it relates to shoulder arthroplasty in an attempt to reduce this bacterial burden prior to surgery. There have been promising results with multi-day preparation skin cleansing with benzoyl peroxide. However, there are no studies looking at intra-operative skin incision preparations targeting the region of skin where the C. acnes bacteria resides. In vitro studies show SURGX antimicrobial gel (Next Science, Jacksonville, FL) results in a marked reduction of C. acnes in addition to other common bacteria affecting prosthetic joints. This gel uses citric acid to chelate the metallic bonds of biofilm. The bacteria are then destroyed by a combination of a high osmolarity environment coupled with a surfactant.

The first purpose of the study is to evaluate if a dermal layer preparation will reduce positive cultures of C. acnes after primary shoulder arthroplasty. There will be a control group consisting of no skin preparation. There will be two additional comparative groups. The second purpose of this study is to compare the use of standard povidone-iodine swab versus SURGX antimicrobial gel as an application into the dermal layer after the skin incision has been made with a skin knife to see if there is a reduction in bacterial burden in the superficial and deep tissues at the end of a primary shoulder arthroplasty. Superficial and deep cultures will be obtained at the conclusion of the shoulder replacement surgery. These cultures will be held in the lab for 2 weeks to identify if bacteria is present. The study team's hypothesis is that the SURGX antimicrobial gel will provide a greater reduction in bacterial burden compared to povidone-iodine within the deep tissues after primary shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned to undergo elective primary anatomic or reverse shoulder arthroplasty.

Exclusion Criteria:

* Patient is undergoing revision shoulder replacement surgery.
* Patient has a known allergy to iodine, benzalkonium chloride, or polythylene glycol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Otto, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by physicians at 1 academic medical center between June 2023 and November 2023.
Pre-assignment Details: 60 participants were enrolled, and all 60 met inclusion criteria and were randomized to a study arm.
Groups:
- No Skin Incision Preparation: The control group will receive no dermal layer skin preparation. At the time of the surgery, after the skin incision has been made with a skin knife, the dermal layer will not be prepped with an agent.
- Povidone-iodine: At the time of the surgery, after the skin incision has been made, the dermal layer will be prepped with povidone-iodine.
  Drug: povidone-iodine Dose: swabstick Administration: swab the incision Frequency: once
  Povidone-Iodine: Applied to skin incision.
- SURGX Wound Gel: At the time of the surgery, after the skin incision has been made, the dermal layer will be prepped with SURGX Wound Gel. SURGX wound gel is a topical antiseptic gel agent to be used on surgical incisions to prevent bacterial infection.
  SURGX Wound Gel: Applied to skin incision.
Period: Overall Study
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.35 (8.443) | 68.50 (10.405) | 68.75 (7.107) | 68.87 (8.615)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 15 | 39
  Male | 10 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 20 | 18 | 56
  Unknown or Not Reported | 2 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 16 | 18 | 18 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.1880 (7.22953) | 32.5010 (5.58499) | 30.7310 (6.53229) | 30.8067 (6.51775)
Type of Shoulder Arthroplasty [Count of Participants; unit: Participants] — Patients included in this study included those undergoing either anatomic total shoulder arthroplasty or reverse total shoulder arthroplasty. These are both shoulder replacement surgeries that involve a different surgical approach.
  Participants
    Reverse TSA | 17 | 19 | 17 | 53
    Anatomic TSA | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Presence of Bacteria Within Shoulder Culture Using Incisional Prep vs. no Prep
Description: Each participant had culture swabs at end of surgical case from deep, superficial, and implant locations. Cultures were held in the lab for 2 weeks to evaluate for the presence of bacteria. The number of patients with at least one positive culture were compared among the three study arms.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel
Number analyzed (Participants) | 20 | 20 | 20
Participants | 11 | 9 | 6
Statistical Analysis 1: Comparison: No Skin Incision Preparation vs Povidone-iodine vs SURGX Wound Gel; Test type: Superiority; p = 0.275, Chi-squared

2. Primary Outcome: Presence of Bacteria Within Shoulder Culture Using Incisional Prep vs. no Prep
Description: Each participant had 5 total culture swabs at end of surgical case from deep (2), superficial (2), and implant (1) locations. Cultures were held in the lab for 2 weeks to evaluate for the presence of bacteria. The number of positive cultures after 2 weeks were compared among the control group and SURGX group.
Time Frame: Day 14
Population: Each participant had 5 total culture swabs at end of shoulder surgery from deep (2), superficial (2), and implant (1) locations.
Measure: Number; unit: # of positive cultures
Units Other Than Participants: culture swabs
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (culture swabs) | 100 | 100 | 100
# of positive cultures | 29 | 24 | 13
Statistical Analysis 1: Comparison: No Skin Incision Preparation vs SURGX Wound Gel; Test type: Superiority; p = 0.0056, Chi-squared

3. Secondary Outcome: Presence of Bacteria Within Shoulder Culture Using SURGX Wound Gel Prep vs. Povidone-iodine Prep
Description: Each participant had culture swabs at end of surgical case from deep, superficial, and implant locations. Cultures were held in the lab for 2 weeks to evaluate for the presence of baceria. The number of patients with at least one positive culture were compared among the SURGX and povidone-iodine groups.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel
Number analyzed (Participants) | 20 | 20 | 20
Participants | 11 | 9 | 6
Statistical Analysis 1: Comparison: Povidone-iodine vs SURGX Wound Gel; Test type: Superiority; p = 0.286, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 weeks after patient surgery through end of study
Description: Adverse events as defined by the protocol were to be collected on the date of patient's surgery and included any type of reaction to the application of product. No follow-up appointments or study procedures after date of surgery are included in this study. The events listed below were considered to be patient complications unrelated to the study, but have been included in this Results section as they meet the clinicaltrials.gov definition of AE.
Arm/Group | No Skin Incision Preparation | Povidone-iodine | SURGX Wound Gel
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 3/20 | 2/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Skin Incision Preparation (N=20) | Povidone-iodine (N=20) | SURGX Wound Gel (N=20)
Infection (Infections and infestations) | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Shoulder dislocation (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Readmission for Social Reasons (Social circumstances) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT05919888/Prot_SAP_000.pdf